CLINICAL TRIAL: NCT07194135
Title: Comparison of Intra-articular Tenoxicam and Triamcinolone Acetonide in the Management of Knee Osteoarthritis: A Randomized Prospective Study
Brief Title: Intra-articular Tenoxicam Versus Triamcinolone Acetonide in Knee Osteoarthritis Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Hossam Mohamed Saad, Lecturer of Orthopedic Surgery, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rc 26-10-2024
Record Dates: First submitted 2025-09-18; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee Osteoarthritis; Intra-articular Injection; Tenoxicam; Non-Steroidal Anti-Inflammatory Drugs; Triamcinolone Acetonide; Corticosteroid Injections; Pain Management
MeSH Terms: conditions — Osteoarthritis, Knee; Agnosia | interventions — tenoxicam; Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a 1:1 ratio to receive either intra-articular tenoxicam or intra-articular triamcinolone acetonide.
Masking Description: This was an open-label trial. Participants and investigators were aware of treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenoxicam Injection (Experimental): Participants received a single intra-articular injection of tenoxicam 20 milligrams, administered aseptically through an anterolateral approach to the knee joint.
  Interventions: Drug: Tenoxicam
- Triamcinolone Acetonide Injection (Active Comparator): Participants received a single intra-articular injection of triamcinolone acetonide 40 milligrams, administered aseptically through an anterolateral approach to the knee joint.
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Tenoxicam — Intra-articular administration of tenoxicam, 20 milligrams as a single injection, delivered through an anterolateral approach under aseptic technique.
  Arms: Tenoxicam Injection
Drug: Triamcinolone Acetonide — Intra-articular administration of triamcinolone acetonide, 40 milligrams as a single injection, delivered through an anterolateral approach under aseptic technique.
  Arms: Triamcinolone Acetonide Injection

SUMMARY:
Knee osteoarthritis is a very common joint condition that leads to pain, stiffness, and difficulty with daily activities, particularly in middle-aged and older adults. Many patients do not get adequate relief from oral pain medications, non-steroidal anti-inflammatory drugs, or physical therapy. Because of this, injections directly into the knee joint are often used.

Corticosteroid medicines, such as triamcinolone acetonide, are among the most frequently used intra-articular injections. They provide strong and rapid anti-inflammatory effects, but their benefits often wear off after only a few weeks. In addition, corticosteroids may cause unwanted systemic effects such as temporary increases in blood sugar, which can be especially concerning for patients with diabetes.

Non-steroidal anti-inflammatory drugs are another group of medicines that can relieve pain and inflammation. Tenoxicam is a long-acting medicine from this group. When given directly into the knee joint, tenoxicam may provide local pain relief for a longer duration, while reducing the amount of drug that circulates in the body. This may lower the risk of side effects compared with oral treatment or repeated corticosteroid injections.

This clinical study was designed to compare the effects of a single intra-articular injection of tenoxicam with a single intra-articular injection of triamcinolone acetonide in patients who have symptomatic knee osteoarthritis. The primary aim was to determine which treatment provides better improvement in knee pain, measured using a visual analog scale. Secondary aims included evaluating knee function using the Western Ontario and McMaster Universities Osteoarthritis Index, monitoring blood sugar control using glycated hemoglobin testing, and assessing the safety of each treatment by recording any local or general adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 45 to 75 years
* Radiographically confirmed knee osteoarthritis (Kellgren-Lawrence grade II-III)
* Persistent knee pain for at least 3 months despite oral non-steroidal anti-inflammatory drugs
* Ability to provide informed consent

Exclusion Criteria:

* Prior intra-articular injection within the past 6 months
* Inflammatory arthritis (e.g., rheumatoid arthritis, gout)
* Advanced knee osteoarthritis (Kellgren-Lawrence grade IV)
* Active joint or systemic infection
* Bleeding disorder or anticoagulant use contraindicating injection
* Uncontrolled diabetes mellitus
* Known hypersensitivity to tenoxicam or triamcinolone acetonide

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-11-03 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Knee Pain Intensity Measured by Visual Analog Scale | Baseline, 2 weeks, 6 weeks, and 12 weeks after injection
  Pain intensity in the affected knee was assessed using a visual analog scale (0 to 100 millimeters), where 0 represents no pain and 100 represents the worst imaginable pain. The outcome was defined as the change from baseline score to follow-up assessments.

SECONDARY OUTCOMES:
Change in Knee Function Measured by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, 2 weeks, 6 weeks, and 12 weeks after injection
  The Western Ontario and McMaster Universities Osteoarthritis Index evaluates pain, stiffness, and physical function in patients with knee osteoarthritis. Scores range from 0 to 96, with higher scores indicating worse symptoms. The outcome was defined as the change from baseline to follow-up.
Change in Glycemic Control Measured by Glycated Hemoglobin (HbA1c) | Baseline and 1 month after injection
  Glycated hemoglobin (HbA1c) was measured to evaluate the effect of intra-articular injection on blood glucose control. The outcome was defined as the change in HbA1c percentage from baseline to one month after injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospitals, Department of Orthopedics and Rheumatology, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in the article will be shared, including baseline characteristics, treatment allocation, outcome measures (visual analog scale for pain, Western Ontario and McMaster Universities Osteoarthritis Index, glycated hemoglobin), and adverse event data. A data dictionary defining each variable will be provided. No directly identifying information will be included.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting documents will be available beginning 6 months after publication of the primary manuscript and for a period of 5 years thereafter.
Access Criteria: Qualified researchers affiliated with an academic or healthcare institution may request access by submitting a brief proposal (study aims, analysis plan, and list of requested variables) and institutional ethics approval or exemption. Access will be granted upon execution of a Data Use Agreement that prohibits re-identification, redistribution, and use beyond the approved proposal. Data will be shared via secure, password-protected transfer or a controlled-access repository designated by the sponsor.